CLINICAL TRIAL: NCT01097005
Title: Special Investigation of Clarith/Klaricid in Patients With Non-tuberculous Mycobacterial Pulmonary Infections
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Collaborators: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: P10-765
Record Dates: First submitted 2010-02-26; First posted 2010-04-01 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2015-03

CONDITIONS: Mycobacterium Infections, Atypical
Keywords: Mycobacterium Infections, Atypical
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Klaricid: Those with an exposure

SUMMARY:
To evaluate the efficacy and safety of long-term treatment with clarithromycin in patients with Non-tuberculous Mycobacterial Pulmonary Infections.

DETAILED DESCRIPTION:
Background: The revised 2007 American Thoracic Society/Infectious Diseases Society of America guidelines recommend a clarithromycin-based combination therapy for treatment of Mycobacterium avium complex (MAC) lung disease and stipulate approximately 1 year of continuous treatment after bacilli negative conversion. However, supporting data are insufficient.

Objectives: To obtain data on the clinical outcome of clarithromycin-based regimens by conducting a nationwide prospective study mainly of MAC lung disease.

Methods: In accordance with the guidelines, patients were enrolled in this survey according to their chest radiographic findings and microbiologic test results. They were treated with a multi-drug regimen including clarithromycin, rifampicin, and ethambutol (clarithromycin -based regimen) until bacilli negative conversion on continual treatment for 1 year. Data were collected "pre-administration," "on the bacilli negative conversion," and "at 6 months after the end of treatment."

ELIGIBILITY:
Inclusion Criteria

* Patients with Pulmonary non-tuberculous mycoplasma infection and who are indicated for treatment with Klaricid

Exclusion Criteria

* Contraindications according to the package insert
* Patients with a history of hypersensitivity to any ingredient of Klaricid
* Patients who are receiving pimozide, ergot-containing products, or cisapride
* Patients who have AIDS (Acquired Immune Deficiency Syndrome)

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pulmonary non-tuberculous mycoplasma infection and who are indicated for treatment with Klaricid
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Kato, MD., Ph.D., Study Director — Abbott Japan Co.,Ltd
Locations (59):
- Japan (59):
  - Site Reference ID/Investigator# 36460, Aichi
  - Site Reference ID/Investigator# 39122, Aichi
  - Site Reference ID/Investigator# 36463, Akita
  - Site Reference ID/Investigator# 36470, Ehime
  - Site Reference ID/Investigator# 36471, Fukuoka
  - Site Reference ID/Investigator# 36472, Fukuoka
  - Site Reference ID/Investigator# 36473, Fukushima
  - Site Reference ID/Investigator# 36474, Gifu
  - Site Reference ID/Investigator# 36475, Hiroshima
  - Site Reference ID/Investigator# 36482, Hyōgo
  - Site Reference ID/Investigator# 36465, Inzai
  - Site Reference ID/Investigator# 36483, Ishikawa
  - Site Reference ID/Investigator# 36484, Kagoshima
  - Site Reference ID/Investigator# 36485, Kanagawa
  - Site Reference ID/Investigator# 36486, Kanagawa
  - Site Reference ID/Investigator# 36487, Kanagawa
  - Site Reference ID/Investigator# 54466, Kitakyushu
  - Site Reference ID/Investigator# 54468, Kobe
  - Site Reference ID/Investigator# 36488, Kochi
  - Site Reference ID/Investigator# 36513, Kofu
  - Site Reference ID/Investigator# 39126, Kumamoto
  - Site Reference ID/Investigator# 36489, Kyoto
  - Site Reference ID/Investigator# 36493, Kyoto
  - Site Reference ID/Investigator# 39123, Kyoto
  - Site Reference ID/Investigator# 54469, Maebashi
  - Site Reference ID/Investigator# 36494, Miyagi
  - Site Reference ID/Investigator# 36495, Miyazaki
  - Site Reference ID/Investigator# 36459, Nagoya
  - Site Reference ID/Investigator# 36461, Nagoya
  - Site Reference ID/Investigator# 54465, Nara
  - Site Reference ID/Investigator# 37145, Obihiro
  - Site Reference ID/Investigator# 36497, Okayama
  - Site Reference ID/Investigator# 39125, Okinawa
  - Site Reference ID/Investigator# 28404, Osaka
  - Site Reference ID/Investigator# 36492, Osaka
  - Site Reference ID/Investigator# 36496, Ōita
  - Site Reference ID/Investigator# 36501, Saitama
  - Site Reference ID/Investigator# 54464, Saitama
  - Site Reference ID/Investigator# 36477, Sapporo
  - Site Reference ID/Investigator# 36478, Sapporo
  - Site Reference ID/Investigator# 36481, Sapporo
  - Site Reference ID/Investigator# 36462, Seto
  - Site Reference ID/Investigator# 36503, Shimane
  - Site Reference ID/Investigator# 36506, Shimotsuke
  - Site Reference ID/Investigator# 36504, Shizuoka
  - Site Reference ID/Investigator# 36505, Shizuoka
  - Site Reference ID/Investigator# 36499, Takatsuki
  - Site Reference ID/Investigator# 15101, Tokyo
  - Site Reference ID/Investigator# 36507, Tokyo
  - Site Reference ID/Investigator# 36508, Tokyo
  - Site Reference ID/Investigator# 36509, Tokyo
  - Site Reference ID/Investigator# 36510, Tokyo
  - Site Reference ID/Investigator# 42710, Tokyo
  - Site Reference ID/Investigator# 54470, Tokyo
  - Site Reference ID/Investigator# 36458, Toyohashi
  - Site Reference ID/Investigator# 36511, Wakayama
  - Site Reference ID/Investigator# 37144, Wakayama
  - Site Reference ID/Investigator# 36512, Yamaguchi
  - Site Reference ID/Investigator# 39124, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Please contact the investigator, and discuss with us.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be registered using a central registration system. The investigators will register eligible patients with the registration center via FAX by 7 days after initiation of clarithromycin treatment.
Groups:
- Clarithromycin: Those with an exposure
Period: Overall Study
Arm/Group | Clarithromycin
Started | 466 (number of participants who were enrolled for this study.)
Analysis of Safety | 441 (number of participants who could be measured for Adverse Events)
Analysis of NTM Lung Disease | 340 (number of participants who contributed to the Baseline data)
Analysis of Bacilli Negative Conversion | 285 (number of participants who were analysed for bacilli negative conversion)
Analysis of CGI | 249 (number of participants who were measured for Clinical Global Improvement (CGI))
Completed | 101
Not Completed | 365
Not completed — Case Report Form not collected | 18
Not completed — Subjects cannot visit the hospital | 1
Not completed — Poor medication compliance | 1
Not completed — No examination data available | 244
Not completed — Deviation from exclusion criteria | 37
Not completed — Adverse Event | 14
Not completed — Discontinuance by complication | 50

BASELINE CHARACTERISTICS:
Arm/Group | Clarithromycin
Number analyzed (Participants) | 340
Age, Customized [Number; unit: participants]
  <45 years | 15
  45-64 years | 136
  65-74 years | 126
  >=75 years | 62
  unknown | 1
Sex/Gender, Customized [Number; unit: participants]
  Female | 256
  Male | 83
  unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Bacilli Negative Conversion Rate
Description: Number of participants who tested positive for Bacilli before treatment and converted to Bacilli Negative at any point during the treatment with clarithromycin
Time Frame: During the treatment with clarithromycin, from 40 days to 1232 days
Population: Analysis of the bacilli negative conversion
Measure: Number; unit: participants
Groups:
- Clarithromycin: Negative conversion / Yes
Arm/Group | Clarithromycin
Number analyzed (Participants) | 285
participants | 269

2. Secondary Outcome: Efficacy Evaluation Using the 4-rank Scale of "Effective", "Ineffective", "Deterioration", or "Impossible" by the Investigator
Description: Number of participants who evaluated for efficacy of clarithromycin with the 4-rank Scales ("Effective", "Ineffective", "Deterioration", "Impossible")
Time Frame: When treatment with clarithromycin is discontinued, from 40 days to 1232 days
Population: Analysis of Clinical Global Improvement (CGI). Number of patients with each rank scale.
Measure: Number; unit: Number of patients
Arm/Group | Clarithromycin
Number analyzed (Participants) | 249
Number of patients
  Effective | 217
  Ineffective | 13
  Deterioration | 10
  Impossible to assess | 9

3. Secondary Outcome: Bacteriological Relapse Related to Duration of Clarithromycin Administration
Description: Number of patients who have bacteriological relapse related to duration of Clarithromycin (CLR) administration after initial negative conversion
Time Frame: 36 months
Population: End of study (completers). Analysis of bacteriological relapse.
Measure: Number; unit: participants
Groups:
- Clarithromycin: The subjects who completed the study
Arm/Group | Clarithromycin
Number analyzed (Participants) | 101
participants
  0-14 months CLR | 5
  ≥15 months CLR | 0

ADVERSE EVENTS:
Time Frame: During treatment with clarithromycin up to 3.4 years
Arm/Group | Clarithromycin
Serious Adverse Events (participants affected / at risk) | 35/441
Other Adverse Events (participants affected / at risk) | 0/441
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clarithromycin (N=441)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Disorientation (Psychiatric disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Somnolence (Nervous system disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causal relationship with the study drug was rated as "possible" by the investigator.
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Weight decreased (Investigations) | 1 (1) — Causal relationship with the study drug was rated as "possible" by the investigator.
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Pneumonia (Infections and infestations) | 3 (3) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Bacterial infection (Infections and infestations) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Pneumonia bacterial (Infections and infestations) | 4 (4) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Atypical mycobacterial infection (Infections and infestations) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Loss of consciousness (Nervous system disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Optic neuritis (Nervous system disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Vertigo positional (Ear and labyrinth disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Arrhythmia (Cardiac disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Cardiac failure acute (Cardiac disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Alveoliltis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Dysphagia (Gastrointestinal disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Large intestine polyp (Gastrointestinal disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Calculus urinary (Renal and urinary disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Haematuria (Renal and urinary disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.
Pyrexia (General disorders) | 1 (1) — Causal relationship with the study drug was rated as "Not related" by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will be granted by sponsor.